CLINICAL TRIAL: NCT05948956
Title: Effects of Combined Exercise Training and Ketone Ester on Muscle Strength and Cardiovascular Response in Parkinson's Disease
Brief Title: Effects of Exercise Training and Ketone Ester on Muscle Strength and Cardiovascular Response in Parkinson's Disease
Acronym: CYCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Chatkaew Pongmala, Research Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00232413
Record Dates: First submitted 2023-06-26; First posted 2023-07-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Exercise; Ketone Ester; Keto
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5-Session Ketone Ester Beverage & Exercise (Experimental): Participants will consume ketone ester (KE) beverage, consisting of 2 scoops (=25 g C8-KE) of Qitone Pro-Ketone Powder™ and electrolyte solution diluted in water, before each of 5 1-hour sessions of aerobic exercise.
  Interventions: Dietary Supplement: Ketone Ester Beverage; Behavioral: Cycling Intervention
- 5-Session Electrolyte Beverage & Exercise (Placebo Comparator): Participants will consume placebo electrolyte (EL) beverage, consisting of an electrolyte solution diluted in water, before each of 5 1-hour sessions of aerobic exercise
  Interventions: Dietary Supplement: Electrolyte Beverage; Behavioral: Cycling Intervention
- 12-Session Ketone Ester Beverage & Exercise (Experimental): Participants will consume ketone ester (KE) beverage, consisting of 2 scoops (=25 g C8-KE) of Qitone Pro-Ketone Powder™ and electrolyte solution diluted in water, before each of 12 1-hour sessions of aerobic exercise.
  Interventions: Dietary Supplement: Ketone Ester Beverage; Behavioral: Cycling Intervention
- 12-Session Electrolyte Beverage & Exercise (Placebo Comparator): Participants will consume placebo electrolyte (EL) beverage, consisting of an electrolyte solution diluted in water, before each of 12 1-hour sessions of aerobic exercise
  Interventions: Dietary Supplement: Electrolyte Beverage; Behavioral: Cycling Intervention

INTERVENTIONS:
Dietary Supplement: Ketone Ester Beverage — Participants will consume ketone ester (KE) beverage, consisting of 2 scoops (=25 g C8-KE) of Qitone Pro-ketone Powder ™ and electrolyte solution diluted in water, before each of 5 or 12 1-hour sessions of aerobic exercise.
  Other Names: Qitone Pro-ketone Powder ™
  Arms: 12-Session Ketone Ester Beverage & Exercise; 5-Session Ketone Ester Beverage & Exercise
Dietary Supplement: Electrolyte Beverage — Participants will consume an electrolyte solution diluted in water, before each of 5 or 12 1-hour sessions of aerobic exercise.
  Arms: 12-Session Electrolyte Beverage & Exercise; 5-Session Electrolyte Beverage & Exercise
Behavioral: Cycling Intervention — Five or twelve 1-hour sessions of cycling on the ergometer over a 2-6 week period. Sessions will consist of a 10 min warm up followed by 8 intervals consisting of 3 min "fast" cycling at 80-90 rpm followed by 2 min of "slow" cycling at ≤60rpm, followed by a 10-minute cool-down.

SUMMARY:
The main purpose of this study is to assess changes in exercise capacity in people with Parkinson's disease before and after an exercise training program with ketone ester supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease

Exclusion Criteria:

* Any recent changes in EKG, history of myocardial infarction or other cardiac event or other cardiac contraindications to exercise
* Inability to use a step, stand, walk, or use a stationary cycle ergometer
* History of symptoms in exercise that preclude safe and comfortable participation, such as dizziness and lightheadedness, orthostasis, severe symptomatic leg or back musculoskeletal pain, painful neuropathy, significant ankle edema or medication side effects
* History of symptomatic cardiovascular or pulmonary disease interfering with exercise
* History of active rheumatoid arthritis
* History of uncontrolled chronic pain syndrome
* Any other history of medical or psychiatric comorbidity precluding safe participation in the project
* Poorly controlled diabetes
* Pregnancy or breastfeeding
* Clinically significant dementia
* Any contraindications to MRI (metal implants, severe claustrophobia, inability to lie still for 1 hour, etc.)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Change in duration of 80 rpm endurance test | After approximately 2-6 weeks of intervention
  Participants will cycle at their personalized fixed wattage at 80 rpm until failure, defined as the point at which the participant could not sustain a cadence of >70 rpm for a cumulative total of 20 s, or until voluntarily choosing to end the test. Change in duration will be calculated by subtracting the baseline duration from duration at follow-up. Greater duration indicates better endurance.
Change in oxygen uptake (VO2 max) | After approximately 2-6 weeks of intervention
  VO2 max (defined as volume of oxygen consumed in mL divided by body weight in kg per minute) will be measured during a controlled cycling session on a stationary bike. Participants will begin at a cadence of 80 rpm at 50 watts for 4 minutes. Thereafter, wattage will increase by 10 watts every 2 minutes until the participant voluntarily ends the session or is no longer able to sustain a cadence of >70 rpm. Participants will wear a face mask that measures their oxygen intake during the session. Change in VO2 max will be calculated by subtracting the baseline VO2 max from VO2 max at follow-up. Greater VO2 max indicates better cardiorespiratory fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Chatkaew Pongmala, PhD, Principal Investigator — University of Michigan
Locations (1):
- Domino's Farms, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT05948956/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT05948956/ICF_001.pdf